CLINICAL TRIAL: NCT00778505
Title: Target-Controlled Infusion of Propofol and Remifentanil During General Anaesthesia Guided by the Index Bispectral: Comparison in Pediatric Patients Between Manual Perfusion and Automated Perfusion
Brief Title: Use of Closed-loop Anesthesia in Pediatric Patients
Acronym: LoopPed
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/21
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia
Keywords: Anesthesia
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): closed-loop administration of propofol and remifentanil using bispectral index as the controller
  Interventions: Drug: Propofol; Drug: remifentanil
- 2 (Active Comparator): manual administration of propofol and remifentanil according to bispectral index values
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Propofol — closed-loop administration using bispectral index as the controller
  Arms: 1
Drug: remifentanil — closed-loop administration using bispectral index as the controller
  Arms: 1
Drug: Propofol — manual administration according bispectral index values
  Arms: 2
Drug: Remifentanil — manual administration according bispectral index values
  Arms: 2

SUMMARY:
To compare manual administration of propofol and remifentanil and dual closed-loop using bispectral index as the control variable during pediatric anesthesia

ELIGIBILITY:
Inclusion Criteria:

* class ASA I, II or III
* general anesthesia scheduled to last more than one hour
* intraoperative hemorrhage planned to be less than 15% of the blood volume

Exclusion Criteria:

* Combined general and regional anesthesia,
* Patients with a pacemaker or scheduled for a cardiac or brain surgical procedure,
* History of a neurological or a psychiatric disorder, or central brain lesion,
* Patients receiving a psychotropic treatment or a a morphine agonist-antagonist,
* Allergy to latex, propofol, remifentanil, morphine, muscle relaxant, or to a component,
* Hypersensibility to remifentanil or to a derivate of fentanyl,
* Scheduled postoperative ventilation or sedation.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of time during which the bispectral index is between 40 and 60 | anesthesia

SECONDARY OUTCOMES:
propofol and remifentanil doses | anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch, Suresnes, France
Locations (2):
- France (2):
  - Hôpital Necker Enfants, Paris
  - Hôpital Foch, Suresnes